CLINICAL TRIAL: NCT05572892
Title: Prognosis Criteria for Walking Independently Recovery After Stroke : Evaluation of the TWIST Algorithm
Brief Title: Prospective Cohort Study : Evaluation of Prognosis Criteria for Walking Independently Recovery After Stroke.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01679-34
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-09

CONDITIONS: Stroke
Keywords: TWIST Algorithm; stroke; prognosis; walking
MeSH Terms: conditions — Stroke | interventions — Thrombin Time; antigens, CD200; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients hospitalised in the Neurology Department of Caen University Hospital: Measurement of walking dependency according to the FAC scale (in the first week after stroke by physiotherapists, at 6 weeks, 12 weeks and 6 months by telephone).
  Interventions: Other: FAC scale

INTERVENTIONS:
Other: FAC scale — Measurement of walking dependency according to the FAC scale :
  * in the first week after stroke (in neurology by physiotherapists),
  * then at 6 weeks, 12 weeks and 6 months (by telephone).
  Trunk Control Test score (in the first week after stroke, by physiotherapists).
  MRC score of hip extension and hip flexion, knee flexion/extension, ankle plantar and dorsal flexion (in the first week after stroke, by physiotherapists).
  PHQ-9 depression scale (at 6 weeks by phone).
  Denutrition (weight loss between neurology weight and 6-week weight, BMI +/- albumin).
  Other intercurrent medical problems (at each telephone interview).
  Other Names: TCT (Trunk Control Test) score; MRC (Medical Research Council) score; PHQ-9 (Patient Health Questionnaire-9) depression scale

SUMMARY:
Based on a 2017 US study that developed an algorithm for predicting independent walking recovery after stroke, we propose a prospective study to assess the validity and applicability of this algorithm in the majority of stroke patients with walking dependence and to confirm its performance.

This study will therefore include adult patients, hospitalised in the Neurology Department of Caen University Hospital, and presenting a dependence on walking according to the FAC (Functional Ambulation Categories) scale in the first week after stroke.

Treated by M. Pierre-Alexis Rousseau (medical intern for Physical and Rehabilitation Medicine), under the direction of Dr. Alexis Ruet, and in collaboration with the physiotherapists of the Neurology Department (Delphine Lebreton and Daphne Scelles), this study is planned to include patients in the initial phase of the stroke, and to continue to follow up the patients until 6 months after their inclusion.

The aim of this work is to evaluate the performance of the TWIST algorithm in predicting walking recovery after stroke according to trunk control (using the Trunk Control Test) and hip extension strength (using the Medical Research Council score), and to analyse other factors that may potentially influence walking recovery (such as visual field amputation, neglect, ataxia, depression, undernutrition).

DETAILED DESCRIPTION:
The ability to walk independently is the most common goal of rehabilitation after a stroke. Whether a patient can walk independently influences decisions about the type and duration of rehabilitation and the proposed destination at discharge from acute care.

The interest of the proposed research is to replicate an American landmark study (The TWIST Algorithm Predicts Time to Walking Independently After Stroke, Smith et al.) published in Neurorehabilitation and Neural Repair in 2017, which developed an algorithm to predict recovery of independent walking after stroke, based on clinical assessment of trunk control by the Trunk Control Test (TCT) and Medical Research Council (MRC) motor strength of hip extension.

The performance of the algorithm in predicting return to walking at 6 and 12 weeks was good (< 6 weeks: Positive Predictive Value = 91%, Negative Predictive Value = 100% // < 12 weeks: Positive Predictive Value = 100%, Negative Predictive Value = 97%), but requires confirmation given the small number of patients included in the study (N = 41).

The originality of the planned research is to try to include and analyse more patients than the original study, to study other factors that may influence recovery, and to continue the follow-up up to 6 months, which wasn't done in the original study.

The expected results would allow the TWIST algorithm to be confirmed in order to better predict walking recovery independently, which could guide rehabilitation and give patients an estimate of their progress towards walking recovery.

The potential benefits for patients would be to maintain motivation for rehabilitation, and to have an impact on the medico-socio-economic level (notably by avoiding investing resources in unlikely objectives).

There are no foreseeable risks, a priori.

If the results are consistent with those of the original study, it may be possible to consider the application of the TWIST algorithm to routine practice for any first stroke causing walking dependence.

Based on the results of the original study, the patients included will be categorised according to their Truck Control Test (TCT) score and their MRC score for hip extension of the deficient limb :

* TCT score > 40 = walking before 6 weeks,
* TCT < 40 + MRC ≥ 3 = walking before 12 weeks,
* TCT < 40 + MRC < 3 = dependent on walking after 12 weeks.

For all included patients: PHQ-9 depression scale and body weight at 6 weeks post-stroke, by telephone.

For patients categorised as " walking before 6 weeks " :

* Call and assessment of FAC scale at 6 weeks,
* If walking (FAC ≥ 4), end of follow-up,
* If not, continuation of follow-up with call at 12 weeks.

For patients categorised as " walking before 12 weeks " :

* Call and assessment of FAC scale at 6 and 12 weeks,
* If walking, end of follow-up,
* If not, continue follow-up with call at 6 months.

For patients categorised as " dependent on walking after 12 weeks " :

- Call and assessment of FAC scale at 6 weeks, 12 weeks and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( ≥ 18 years) hospitalised in the Neurology Department of Caen University Hospital
* FAC scale score < 4 (walking dependent) in the first week after stroke
* Oral and written comprehension of the French language
* Affiliation to a social security scheme

Exclusion Criteria:

* Patient dependent on walking (FAC < 4) before stroke
* Short-term (< 3 months) life-threatening condition
* Communication impairment (severe aphasia, impaired consciousness) and/or cognitive impairment preventing informed consent and/or rehabilitation
* Opposition of the patient
* Patient under legal protection (guardianship or curators)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients ( ≥ 18 years) hospitalised in the Neurology Department of Caen University Hospital who present stroke with walking dependance (FAC scale score < 4)
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Categories (FAC) | Change from Baseline (first week after stroke) FAC score at 6 weeks after stroke
  Functional Ambulation Categories (FAC) to classify the patient's walking as dependent or non-dependent.
Functional Ambulation Categories (FAC) | Change from Baseline (1 week after stroke) FAC score at 12 weeks after stroke
  Functional Ambulation Categories (FAC) to classify the patient's walking as dependent or non-dependent.

SECONDARY OUTCOMES:
Age | At first week after stroke
  Demographic characteristic
Gender | At first week after stroke
  Demographic characteristic
National Institutes of Health Stroke Scale (NIHSS) score | At first week after stroke
  Clinical characteristic
"Visual field" item of the National Institutes of Health Stroke Scale (NIHSS)score | At first week after stroke
  Clinical characteristic
"Extinction and neglect" item of the National Institutes of Health Stroke Scale (NIHSS)score | At first week after stroke
  Clinical characteristic
"Ataxia" item of the National Institutes of Health Stroke Scale (NIHSS)score | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC) score for hip extension | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC)score for hip flexion | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC)score for knee extension | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC)score for knee flexion | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC)score for ankle plantar flexion | At first week after stroke
  Clinical characteristic
Medical Research Council (MRC)score for ankle dorsal flexion | At first week after stroke
  Clinical characteristic
Patient Health Questionnaire (PHQ-9) depression scale | At 6 weeks after stroke
  Description of the patient's mental health status at the end of the PHQ-9 depression questionnaire
Undernutrition | At 6 weeks after stroke
  Search for weight loss between the weight in neurology and the weight at 6 weeks, Body Mass Index +/- albumin

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ruet, Study Director — Physical Medicine and Rehabilitation Department in the University Hospital of Caen; Pierre Alexis Rousseau, Principal Investigator — Physical Medicine and Rehabilitation Department in the University Hospital of Caen; Clemence Tomadesso, Study Chair — Clinical Research Unit of University Hospital of Caen
Locations (1):
- University Hospital of Caen Normandie, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith MC, Barber PA, Stinear CM. The TWIST Algorithm Predicts Time to Walking Independently After Stroke. Neurorehabil Neural Repair. 2017 Oct-Nov;31(10-11):955-964. doi: 10.1177/1545968317736820. Epub 2017 Nov 1. PMID 29090654
- [Background] Williams LS, Brizendine EJ, Plue L, Bakas T, Tu W, Hendrie H, Kroenke K. Performance of the PHQ-9 as a screening tool for depression after stroke. Stroke. 2005 Mar;36(3):635-8. doi: 10.1161/01.STR.0000155688.18207.33. Epub 2005 Jan 27. PMID 15677576